CLINICAL TRIAL: NCT03477331
Title: Antithrombotics' Therapeutic Optimization in Hospitalized Patients Using Physiologically- and Population-based Pharmacokinetic Modeling
Acronym: OptimAT
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Jean-Luc Reny, Prof, University Hospital, Geneva
Other Study IDs: 2017-00225
Record Dates: First submitted 2018-02-02; First posted 2018-03-26 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Cardiovascular Diseases
Keywords: Direct oral anticoagulant; P2Y12 inhibitors; Physiologically-based pharmacokinetic model (PBPK); Population-based pharmacokinetic model (POPPK)
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main goal of the OptimAT study main goal is to validate a PBPK model for 3 direct oral anticoagulants (rivaroxaban, apixaban, dabigatran) and 3 P2Y12 inhibitors (clopidogrel, ticagrelor, prasugrel) in hospitalized patients.

DETAILED DESCRIPTION:
Patients treated with antithrombotics are at risk of both severe ischemic and bleeding events. However, current clinical scores are insufficiently discriminant to predict the most favorable drug and dosing for an improved net clinical benefit. Physiologically and population-based pharmacokinetic models (PBPK and POPPK respectively) incorporate substrate specific properties obtained from experimental in-vitro experiments as well as patients' demographic, genetic and physiological in vivo data in order to characterize the dose-concentration relationships. As such, they can be used to simulate and predict PK profiles accounting for specific patients' characteristics and are the basis of dosing optimization. These models could be a valuable tool to predict antithrombotic blood concentration in a given patient. Our main goal is to elaborate predictive models characterizing the dose-concentration relationship with influencing variables of three direct oral anticoagulants (DOAC) (rivaroxaban, apixaban, dabigatran) and three P2Y12 inhibitors (clopidogrel, prasugrel, ticagrelor) in hospitalized patients, which will serve as basis for drug selection and dosage optimization.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients at any of the Geneva University Hospitals 18 yo and older
* Treated with DOAC (dabigatran, rivaroxaban, apixaban) or/and P2Y12 (clopidogrel, ticragrelor et prasugel) at the time of study blood sampling
* Understanding of French language and able to give an inform consent.

Exclusion Criteria:

* Patients with a reduced life span (<6 mois)
* Exclusion criteria during follow up
* Change in dosage or cessation of the DOAC or P2Y12 taken by the participant follow up data will be censored at the time of change.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients
Sampling Method: Probability Sample
Enrollment: 444 (Actual)
Dates: Start 2018-01-14 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) | 2 years
  Difference between observed and PBPK model-predicted AUC (mean prediction error)

SECONDARY OUTCOMES:
Trough Concentration (Cmin) | 2 years
  Difference between observed and PBPK model-predicted Cmin (mean prediction error)
Area Under the Curve (AUC) (stability of the model over time) | 2 years
  Difference between observed and model-predicted AUC during patients' rehospitalization (stability of the model over time)
Major bleeding event-free survival | 2 years
  Major bleeding event-free survival according to drug exposure (AUC) during a prospective during a follow-up of two years for DOACs (dabigatran, rivaroxaban, apixaban) and P2Y12 receptor inhibitors (clopidogrel, ticragrelor, prasugel)
Peak concentration (Cmax) | 2 years
  Difference between observed and PBPK model-predicted Cmax (mean prediction error)
Thrombosis event-free survival | 2 years
  Thrombosis event-free survival according to drug exposure (AUC) during a prospective during a follow-up of two years for DOACs (dabigatran, rivaroxaban, apixaban) and P2Y12 receptor inhibitors (clopidogrel, ticragrelor, prasugel)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Reny, Prof, Principal Investigator — University Hospital, Geneva
Locations (1):
- Hopitaux universitaires de Genève, 4 rue Gabrielle-Perret-Gentil, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Terrier J, Gaspar F, Gosselin P, Raboud O, Lenoir C, Rollason V, Csajka C, Samer C, Fontana P, Daali Y, Reny JL; OptimAT study group. Apixaban and rivaroxaban's physiologically-based pharmacokinetic model validation in hospitalized patients: A first step for larger use of a priori modeling approach at bed side. CPT Pharmacometrics Syst Pharmacol. 2023 Dec;12(12):1872-1883. doi: 10.1002/psp4.13036. Epub 2023 Oct 4. PMID 37794718
- [Background] Gaspar F, Terrier J, Favre S, Gosselin P, Fontana P, Daali Y, Lenoir C, Samer CF, Rollason V, Reny JL, Csajka C, Guidi M. Population pharmacokinetics of apixaban in a real-life hospitalized population from the OptimAT study. CPT Pharmacometrics Syst Pharmacol. 2023 Oct;12(10):1541-1552. doi: 10.1002/psp4.13032. Epub 2023 Sep 18. PMID 37723920
- [Background] Achour B, Gosselin P, Terrier J, Gloor Y, Al-Majdoub ZM, Polasek TM, Daali Y, Rostami-Hodjegan A, Reny JL. Liquid Biopsy for Patient Characterization in Cardiovascular Disease: Verification against Markers of Cytochrome P450 and P-Glycoprotein Activities. Clin Pharmacol Ther. 2022 Jun;111(6):1268-1277. doi: 10.1002/cpt.2576. Epub 2022 Mar 28. PMID 35262906
- [Derived] Gaspar F, Jacost-Descombes C, Gosselin P, Reny JL, Guidi M, Csajka C, Samer C, Daali Y, Terrier J. Improving Understanding of Fexofenadine Pharmacokinetics to Assess Pgp Phenotypic Activity in Older Adult Patients Using Population Pharmacokinetic Modeling. Clin Pharmacokinet. 2025 Feb;64(2):275-283. doi: 10.1007/s40262-024-01470-4. Epub 2025 Jan 11. PMID 39798016
- See also: Liquid Biopsy for Patient Characterization in Cardiovascular Disease: Verification against Markers of Cytochrome P450 and P-Glycoprotein Activities — http://ascpt.onlinelibrary.wiley.com/doi/10.1002/cpt.2576